CLINICAL TRIAL: NCT02808299
Title: Liver Injury by Statins in Coronary Heart Disease (CHD) Patients With History of Hepatitis B Virus (HBV) Infection
Brief Title: Liver Injury by Statins in Patients With History of Hepatitis B Virus Infection
Acronym: LISHBV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: StatinsHBV-1
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Liver Injury; Hepatitis B Virus Infection History
Keywords: statin; hepatitis B virus
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- all the antigen and antibody of HBV are negative: Hepatitis B Virus surface antigen (HBsAg), Hepatitis B Virus surface antibody (HBsAb), Hepatitis B Virus e antigen (HBeAg), Hepatitis B Virus e antibody (HBeAb), Hepatitis B Virus core antibody (HBcAb) are all negative.
- HBV infection history: One or more of HBsAb,HBeAb, HBcAb are positive, while HBsAg and HBeAg are negative. If only HBsAb is positive, the history of HBV vaccination need to be excluded.
  Interventions: Other: HBV infection history
- HBV carriers: One or two of HBsAg and HBeAg are positive, accompanied by any HBV antibody is positive or not.
  Interventions: Other: HBV infection history

INTERVENTIONS:
Other: HBV infection history — HBV infection history or HBV carriers
  Other Names: HBV carriers
  Groups: HBV carriers; HBV infection history

SUMMARY:
The purpose of this study is to investigate the incidence of liver injury by statins in coronary heart disease (CHD) patients with history of hepatitis B virus (HBV) infection.

ELIGIBILITY:
Inclusion Criteria:

* patients with CHD receive long-term statin treatment

Exclusion Criteria:

* ALT is over ULN at baseline
* infection of Hepatitis A Virus, Hepatitis C Virus or Hepatitis E Virus
* triglyceride is over 4.5 mmol/L
* decompensated liver cirrhosis (Child B or C)
* active stage of HBV
* infection of Burkitt's lymphoma virus or cytomegalovirus, or other acute infectious disease
* congestive heart failure
* malignant tumor
* autoimmune disease
* receive other potential hepatotoxicity drugs such as immunosuppressant, antituberculotic and non-steroid anti-inflammatory drug.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosied as coronary heart disease (CHD) at hospitalization receive long-term statin treatment, with or without HBV infection history.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
changes of alanine transaminase (ALT, U/L) | one month, three months, six months
  The peak increases of ALT from baseline to follow-up
number of participants with alanine transaminase (ALT) increasing over 3 folds of upper limit normally (ULN) | one month, three months, six months

SECONDARY OUTCOMES:
number of participants with alanine transaminase (ALT) increasing over the ULN | one month, three months, six months

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Yang, Doctor, Study Chair — First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Bellosta S, Paoletti R, Corsini A. Safety of statins: focus on clinical pharmacokinetics and drug interactions. Circulation. 2004 Jun 15;109(23 Suppl 1):III50-7. doi: 10.1161/01.CIR.0000131519.15067.1f. PMID 15198967
- [Background] Ekstedt M, Franzen LE, Mathiesen UL, Holmqvist M, Bodemar G, Kechagias S. Statins in non-alcoholic fatty liver disease and chronically elevated liver enzymes: a histopathological follow-up study. J Hepatol. 2007 Jul;47(1):135-41. doi: 10.1016/j.jhep.2007.02.013. Epub 2007 Mar 8. PMID 17400325
- [Background] Segarra-Newnham M, Parra D, Martin-Cooper EM. Effectiveness and hepatotoxicity of statins in men seropositive for hepatitis C virus. Pharmacotherapy. 2007 Jun;27(6):845-51. doi: 10.1592/phco.27.6.845. PMID 17542767
- [Background] Balmer ML, Dufour JF. Treatment of hypercholesterolemia in patients with primary biliary cirrhosis might be more beneficial than indicated. Swiss Med Wkly. 2008 Jul 26;138(29-30):415-9. doi: 10.4414/smw.2008.12311. PMID 18654866
- [Background] Cohen DE, Anania FA, Chalasani N; National Lipid Association Statin Safety Task Force Liver Expert Panel. An assessment of statin safety by hepatologists. Am J Cardiol. 2006 Apr 17;97(8A):77C-81C. doi: 10.1016/j.amjcard.2005.12.014. Epub 2006 Feb 3. PMID 16581333
- [Background] Watkins PB, Seeff LB. Drug-induced liver injury: summary of a single topic clinical research conference. Hepatology. 2006 Mar;43(3):618-31. doi: 10.1002/hep.21095. PMID 16496329
- [Background] Lu J, Zhou Y, Lin X, Jiang Y, Tian R, Zhang Y, Wu J, Zhang F, Zhang Y, Wang Y, Bi S. General epidemiological parameters of viral hepatitis A, B, C, and E in six regions of China: a cross-sectional study in 2007. PLoS One. 2009 Dec 24;4(12):e8467. doi: 10.1371/journal.pone.0008467. PMID 20041146
- [Result] Zhang Q, Yang Z. Can statins be used safely in coronary heart disease patients of hepatitis B virus carriers? Int J Cardiol. 2011 Jan 21;146(2):291. doi: 10.1016/j.ijcard.2010.10.087. Epub 2010 Dec 3. No abstract available. PMID 21129795
- See also: Click here for more information about this study — http://onlinelibrary.wiley.com/doi/10.1592/phco.27.6.845/abstract;jsessionid=D7FEEA8665D404AD4218069CD7F718D2.f01t01
- See also: Click here for more information about this study — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2794385/